CLINICAL TRIAL: NCT04668131
Title: Study on Curative Effect and Mechanism of Acupuncture on Neuropathic Pain in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200922
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye
Keywords: dry eye; pain; acupuncture
MeSH Terms: conditions — Dry Eye Syndromes; Pain | interventions — Lubricant Eye Drops; Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial tears (Experimental): Artificial tears
  Interventions: Drug: Sodium hyaluronate eye drops
- Acupuncture (Active Comparator): Acupuncture
  Interventions: Other: acupuncture

INTERVENTIONS:
Drug: Sodium hyaluronate eye drops — eye drops, three times a day
  Other Names: artificial tears
  Arms: Artificial tears
Other: acupuncture — three times a week
  Arms: Acupuncture

SUMMARY:
This project is designed as a prospective, randomized, open, controlled clinical trial. For the first time, acupuncture was applied to the treatment of dry ocular neuropathic pain. Its mechanism was discussed by comparing the efficacy between acupuncture and artificial tears.

ELIGIBILITY:
Inclusion Criteria:

* According to the DEWS diagnostic criteria, the OSDI score ≥ 13, with positive signs of dry eye (SIt ≤ 10mm/5min or TBUT ≤ 10s) or CFS positive;
* VAS>0;
* Signed informed consent.

Exclusion Criteria:

* Patients with dry eye who have had irritants directly irritating the ocular surface in the past 3 days;
* Eyeball infections, allergies, deformities, abnormal movements
* Any history of eye surgery
* Have had eye trauma or fundus laser treatment within 3 months
* Used drugs that affect tear production such as antihistamines, antidepressants, etc. within 30 days
* Suffer from systemic diseases that affect tear production, including Sjogren's syndrome, diabetes, mental illness, malignant tumors, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Score | The treatment period for each enrolled subject is one month
  Ask the patient to mark the corresponding position on the ruler that can represent the pain or discomfort during the onset

SECONDARY OUTCOMES:
OSDI | The treatment period for each enrolled subject is one month
  OSDI consists of 12 scoring items, divided into three parts: severity of symptoms, impact of symptoms on daily life, and impact of environment on symptoms.
TBUT | The treatment period for each enrolled subject is one month
  Drop 1 drop of 0.3% sodium fluorescein eye solution into the subject's conjunctival sac, dry it with a sterile cotton swab, and ask him to blink gently to make the fluorescein sodium evenly distributed. Observe the subject from the last time with a slit lamp cobalt blue light. The time from blinking to the first dark spot on the corneal surface, record three times and take the average
SIt | The treatment period for each enrolled subject is one month
  Fold one end of the special 5mm×35mm filter paper (Tianjin Jingming) for tears by 5mm, and gently place it on the middle and outer 1/3 of the subject's lower eyelid conjunctival sac, and the other end will droop naturally. Ask the subject to gently close their eyes for 5 minutes After measuring the length of the filter paper wetted by tears
CFS score | The treatment period for each enrolled subject is one month
  Divide the cornea into 5 quadrants (central + nose/temporal/upper/lower), each quadrant has a staining score of 0 to 3 points, and it is specified that no staining is 0 points, and 30 spots are stained as 1 point, and there is flaky staining and fusion 3 points for filament formation, 2 points between the two, the sum of 5 quadrants is the score of the entire cornea, and the CFS score of the entire cornea is 0-15 points.
Density and curvature of corneal subbasal nerve | The treatment period for each enrolled subject is one month
  Collect corneal subbasal nerve images, 2 images each in the upper, lower, arm, temporal and central areas. Use deep learning methods to analyze nerve density and curvature
Tear pain factor content | The treatment period for each enrolled subject is one month
  With the aid of a slit lamp, a capillary pipette was used to draw 5 μl tears/eye at the middle and outer edges of the lower eyelid 2/3 of the tear river, and placed in a low protein adhesion EP tube (containing 5 μl 1% BSA) and stored at -80°C. ELISA analyzes the protein levels of PGE2, substance P and NGF in tear fluid.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No